CLINICAL TRIAL: NCT00850824
Title: Diabetes Care in American Samoa
Brief Title: Community Health Workers in Diabetes Care in American Samoa
Acronym: DCAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Brown University (Other); The Miriam Hospital (Other); Tafuna Family Health Center (Unknown)
Responsible Party: Principal Investigator, Stephen McGarvey, Professor of Epidemiology and Anthropology, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R18 DK075371-DCAS; NIH Grant R18-DK075371; R18DK075371 (NIH)
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2015-10-07 (Estimated); Status verified 2015-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: T2DM
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Behavioral (Experimental): Community Health Worker home visits
  Interventions: Behavioral: Community Health Worker home visits
- Usual Care (Active Comparator): Usual Care, Wait List Control
  Interventions: Behavioral: Community Health Worker home visits

INTERVENTIONS:
Behavioral: Community Health Worker home visits — Community health workers will educate diabetes patients and families about need for regular medical care, taking medications, increasing exercise patterns, improving diet, keeping medical referral exams for specialty.

SUMMARY:
As type 2 diabetes prevalence increases in the United States, the burden of diabetes falls more on groups with greater barriers to care, such as language and cultural differences, and lower economic resources. Healthy People 2010 targeted diabetes as one of six diseases for the elimination of racial and ethnic health disparities. These disparities extend to the US Territory of American Samoa, where the proportion of adults >18 years with diabetes was 19.6% in 2002, compared to 6.4% of US adults. There have been no reported diabetes interventions in Samoans in the US. The overall purpose of this application is to translate recent advances in diabetes care into clinical practice for the American Samoan community by improving methods of health care delivery and methods of diabetes self management. We will conduct a randomized clinical trial to test the effectiveness of a community health worker (CHW) and primary-care coordinated intervention to provide outreach, education and support to 352 type 2 diabetes patients and their families in American Samoa. The CHW intervention will utilize evidence-based algorithms and protocols to prompt risk behavior interventions, communication with health care team, and visit schedule. The individual treatment action plans are also guided by the Precede-Proceed Model. The outcomes at a one-year follow-up will include glycosolated hemoglobin (HbA1c), cardiovascular disease risk factors, diet and exercise behaviors, and adherence to diabetes care guidelines. The study hypothesis is that diabetes patients in the CHW trial arm will have lower HbA1c levels, lower cardiovascular disease risk factor levels, increased exercise behaviors and healthy dietary intakes and greater adherence to diabetes care such as adherence to prescribed medications, keeping medical appointments for diabetes care and specialty referrals. The intervention builds upon best clinical practices for CHWs in diabetes care by translating effective strategies to American Samoans, while also extending prior CHW research, by using a model that is potentially replicable in other ethnic minority populations suffering the burden of diabetes.

DETAILED DESCRIPTION:
We will perform a clinical trial to test the effectiveness of a community health worker (CHW) and primary-care coordinated intervention to provide outreach, education and support to diabetes patients and their families. The outcomes at a one-year follow-up will include glycosolated hemoglobin (HbA1c), CVD risk factors, diet and exercise behaviors, and adherence to diabetes care guidelines. The intervention builds upon best practices to date with CHWs, by translating effective strategies to Samoans, an ethnic minority population with no prior intervention research, while also extending prior CHW research, by using a model that is potentially replicable anywhere that uses outreach strategies in the context of primary care. This application builds on the current more limited activities of CHWs at the Tafuna Family Health Center (TFHC), a primary care health center established in 1998, operated by the American Samoa Government Department of Health, and designated as a community health center by the U.S. Bureau of Primary Health Care in 2003.

We will conduct a randomized controlled trial to test the effectiveness of a CHW outreach intervention, compared to usual care (UC) in a wait-list control group. The specific aims are:

A.1. To improve control of diabetes: We hypothesize that the CHW outreach intervention group will have greater one-year reductions in glycosolated hemoglobin (HbA1c) levels compared to the UC group.

A.2. To improve cardiovascular risk factors: We hypothesize that the CHW outreach intervention group will have greater one-year reductions in systolic and diastolic blood pressure, BMI, and abdominal circumference compared to the UC Group.

A.3. To improve diet and physical activity behaviors: We hypothesize that the diabetes patients randomized to the CHW intervention will have a greater one-year increase in favorable dietary and physical activity behaviors associated with self-management of their diabetes compared to the UC group.

A.4. To improve adherence to processes of diabetes care. The CHW group will have a higher percent of diabetes patients with the following American Diabetes Association (ADA) standards of care: 1) at least two HBA1c tests in the last year (at least 3 months apart), 2) percent of patients with documentation of self-management goals in the past 12 months, 3) percent of patients with a dental exam in past year, 4) percent of patients with a dilated eye exam in the past year, 5) percent of patients with a documented foot exam in the past year. We hypothesize that the CHW intervention will outperform UC on these variables over one year.

ELIGIBILITY:
Inclusion Criteria: diagnosis of type 2 diabetes, age 21 years and above, resident of American Samoa receiving primary care at Tafuna Family Health Center -

Exclusion Criteria: pregnancy, receiving kidney dialysis

-

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2007-10; Primary Completion 2011-06 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
glycosolated hemoglobin (HbA1c) levels | one year

SECONDARY OUTCOMES:
Blood pressure | one year
serum lipid levels | one year
abdominal circumference | one year
changes in exericse patterns | one year
changes in dietary intake | one year
keeping scheduled medical appointments | one year
keeping specialty referral for medical exams | one year

CONTACTS AND LOCATIONS:
Overall Officials: Stephen T McGarvey, PhD, MPH, Principal Investigator — Brown University, Providence, RI, USA
Locations (1):
- Tafuna Family Health Center, Pago Pago, American Samoa

REFERENCES:
- [Background] Elstad E, Tusiofo C, Rosen RK, McGarvey ST. Living with Ma'i Suka: individual, familial, cultural, and environmental stress among patients with type 2 diabetes mellitus and their caregivers in American Samoa. Prev Chronic Dis. 2008 Jul;5(3):A79. Epub 2008 Jun 15. PMID 18558029
- [Background] Rosen RK, DePue J, McGarvey ST. Overweight and diabetes in American Samoa: the cultural translation of research into health care practice. Med Health R I. 2008 Dec;91(12):372-3, 376-7. No abstract available. PMID 19170313
- [Background] DePue JD, Rosen RK, Batts-Turner M, Bereolos N, House M, Held RF, Nu'usolia O, Tuitele J, Goldstein MG, McGarvey ST. Cultural translation of interventions: diabetes care in American Samoa. Am J Public Health. 2010 Nov;100(11):2085-93. doi: 10.2105/AJPH.2009.170134. Epub 2010 Sep 23. PMID 20864729
- [Background] Held RF, DePue J, Rosen R, Bereolos N, Nu'usolia O, Tuitele J, Goldstein M, House M, McGarvey S. Patient and health care provider views of depressive symptoms and diabetes in American Samoa. Cultur Divers Ethnic Minor Psychol. 2010 Oct;16(4):461-7. doi: 10.1037/a0020089. PMID 21058808
- [Background] Stewart DW, Depue J, Rosen RK, Bereolos N, Goldstein MG, Tuitele J, Nu'usolia O, McGarvey ST. Medication-taking beliefs and diabetes in American Samoa: a qualitative inquiry. Transl Behav Med. 2013 Mar 1;3(1):30-38. doi: 10.1007/s13142-012-0114-y. Epub 2012 Feb 1. PMID 23539136
- [Result] DePue JD, Dunsiger S, Seiden AD, Blume J, Rosen RK, Goldstein MG, Nu'usolia O, Tuitele J, McGarvey ST. Nurse-community health worker team improves diabetes care in American Samoa: results of a randomized controlled trial. Diabetes Care. 2013 Jul;36(7):1947-53. doi: 10.2337/dc12-1969. Epub 2013 Feb 7. PMID 23393217
- [Result] DePue JD, Rosen RK, Seiden A, Bereolos N, Chima ML, Goldstein MG, Nu'usolia O, Tuitele J, McGarvey ST. Implementation of a culturally tailored diabetes intervention with community health workers in American Samoa. Diabetes Educ. 2013 Nov-Dec;39(6):761-71. doi: 10.1177/0145721713504630. Epub 2013 Sep 19. PMID 24052204
- [Result] Hamid S, Dunsiger S, Seiden A, Nu'usolia O, Tuitele J, DePue JD, McGarvey ST. Impact of a diabetes control and management intervention on health care utilization in American Samoa. Chronic Illn. 2014 Jun;10(2):122-34. doi: 10.1177/1742395313502367. Epub 2013 Oct 1. PMID 24085749
- [Derived] Huang SJ, Galarraga O, Smith KA, Fuimaono S, McGarvey ST. Cost-effectiveness analysis of a cluster-randomized, culturally tailored, community health worker home-visiting diabetes intervention versus standard care in American Samoa. Hum Resour Health. 2019 Mar 5;17(1):17. doi: 10.1186/s12960-019-0356-6. PMID 30836964
- [Derived] Rao M, DePue JD, Dunsiger S, Elsayed M, Nu'usolia O, McGarvey ST. Long-Term Impact of a Community Health Worker Intervention on Diabetes Control in American Samoa. Prev Chronic Dis. 2015 Oct 22;12:E180. doi: 10.5888/pcd12.150160. PMID 26491815